CLINICAL TRIAL: NCT02347891
Title: Belimumab for Maintenance Therapy in Idiopathic Inflammatory Myositis
Brief Title: Belimumab in Idiopathic Inflammatory Myositis
Acronym: BIM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Galina Marder, MD, Director, Inflammatory Muscle Disease and Vasculitis Center, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-621
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Myositis
Keywords: Inflammatory Myositis; Dermatomyositis; Polymyositis; Muscle Pain; Myositis; Refractory myositis
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis; Myalgia | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Belimumab + Standard of Care (Experimental): Patients in this arm will be given belimumab with a background of standard of care therapy during the randomized controlled treatment period.
  Patients in this arm will continue to receive belimumab during the open label phase of the study (week 40 - week 64)
  Interventions: Drug: Belimumab
- Placebo + Standard of Care (Active Comparator): Patients in this arm will be given a placebo with a background of standard of care therapy during the randomized controlled treatment period.
  Patients in this arm will receive belimumab during the open label phase of the study (week 40 - week 64).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belimumab — Randomized phase: Week 0 - Week 40
  Other Names: Benlysta
  Arms: Belimumab + Standard of Care
Drug: Placebo — Randomized phase: Week 0 - Week 40
  Other Names: Saline IV bag
  Arms: Placebo + Standard of Care

SUMMARY:
The goal of the trial is to evaluate the efficacy and safety of belimumab as a maintenance therapy in adults with refractory Idiopathic inflammatory myositis (IIM) as compared with standard of care. This is a multicentre double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Adults with refractory IIM will be enrolled. IIM is defined as Dermatomyositis (DM) or Polymyositis (PM), meeting the Bohan & Peter (1975) diagnostic criteria for definite or probable DM or PM. Refractory IIM is defined as chronic active IIM with a history of inadequate response or intolerance to three months of glucocorticoids and/or at least a history of inadequate response or intolerance to three months of one other immunosuppressive agent (IS) (azathioprine, methotrexate, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine, cyclophosphamide, Rituximab or intravenous gamma globulin [IVIG]).

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the study must meet the following inclusion criteria:

1. Adults >18 years of age
2. Have a diagnosis of:

   1. definite or probable dermatomyositis (DM) or
   2. Definite or probable diagnosis of polymyositis (PM) with presence of one of myositis specific antibodies. In the absence of myositis specific auto-antibodies, the diagnosis of PM will require review of the muscle biopsy and adjudication by the predetermined committee of experts.
3. Presence of positive autoantibody (ANA >1:80 or RNP or SSA/SSB or any of the myositis specific autoantibody: antisynthetase autoantibodies (anti-Jo-1, PL-7, PL-12, EJ, OJ, KS), anti-SRP, anti-Mi-2, anti-p140).
4. Have refractory IIM as defined by inadequate response or intolerance to at least 3 months of glucocorticoids and/or at least one other immunosuppressive agent, such as azathioprine, methotrexate, IVIG, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine cyclophosphamide, and Rituximab.
5. Have active IIM at screening. This requires at least 3 criteria from the CSM
6. Dermatomyositis patients that do not meet the MMT criteria, must have:

   1. a cutaneous VAS score of >3 cm on a 10 cm VAS scale (MDAAT) will be required:
   2. elevation of at least one muscle enzyme (creatine kinase [CK]; aldolase; lactate dehydrogenase [LDH]; alanine aminotransferase [ALT]; or aspartate aminotransferase [AST]) to a minimum level of 1.3 times the upper limit of normal,
   3. and 1 additional core set measure
7. For patients with ≥ 7 years of IIM, muscle biopsy or muscle MRI within 4 months prior to enrollment will be required to document active myositis to avoid enrolling patients with significant index of damage/ muscle atrophy. This is not applicable to DM patients with a cutaneous VAS score of >3 cm on a 10 cm VAS scale (MDAAT).
8. Have a stable background glucocorticoid therapy for at least 2 weeks prior to screening (Prednisone (or equivalent) dose < 15 mg daily)
9. Have a stable immunosuppressive therapy (IS) (azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine for > 2 months prior to screening. Patients on intravenous gamma globulin (IVIG) have to be on a stable dose and frequency regimen for ≥ 3 months.
10. Have the ability to understand the requirements of the study and provide written informed consent (including consent for the use and disclosure of research-related health information) and comply with the study protocol procedures (including required study visits)
11. Female subjects of childbearing potential must have a negative urine pregnancy test at screening and agree to 1 of the following:

    1. Complete abstinence from intercourse from 2 weeks prior to administration of the 1st dose of study agent until 16 weeks after the last dose of study agent (Sexual inactivity by abstinence must be consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception); or
    2. Consistent and correct use of 2 of acceptable methods of birth control for 1 month prior to the start of the study agent, during the study, and 16 weeks after the last dose of study agent

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Have severe muscle damage as defined by a Muscle Damage Index (MDI) > 5.0 cm using a visual analogue scale (VAS) 10.0 cm in length or evidence of severe muscle atrophy on muscle MRI.
2. History of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell).
3. Have a history of a primary immunodeficiency
4. Have a significant IgG deficiency (IgG level < 400 mg/dl) Have an IgA deficiency (IgA level < 10 mg/dL)
5. Discontinuation IS agent < 3 months prior to Screening. Including: azathioprine, methotrexate, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine, or intravenous gamma globulin [IVIG]
6. Have received Rituximab within 365 days prior to Screening.
7. Have received cyclophosphamide within 180 days prior to Screening
8. Have received treatment with:

   1. Initiated IVIG 3 months prior to Screening
   2. Pulse steroids 2 months prior to Screening
9. Have received treatment with Belimumab at any time prior to Screening
10. Have received a biologic investigational agent within 365 days prior to Screening.
11. Have received a non-biologic investigational agent within 30 days or 5 half-lives of the agent (whichever is longer) prior to Screening.
12. Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
13. Infection history:

    1. Currently on any suppressive therapy for a chronic infection (such as tuberculosis - including latent tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).

       NOTE: Testing for latent TB is a standard of care for patients on immunosuppressive therapy and results will be obtained from their medical record. If no TB history is found for these patients, a Quantiferon Gold or PPD test will be performed prior to Day 0 as part of standard of care.
    2. Hospitalization for treatment of infection within 60 days of Day 0.
    3. Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 60 days of Day 0.
14. Have a historically positive HIV test or test positive at screening for HIV.
15. Have a history of autoimmune hepatitis
16. Hepatitis status will be obtained from patients' medical records. If unavailable, testing will be done as part of standard of care. Patients are excluded if there is evidence of infection with:

    a. Hepatitis B: i. Positive hepatitis B surface antigen (HBsAg) or positive hepatitis B core antibody (HBcAb) or b. Hepatitis C: i. Positive hepatitis C antibody with confirmatory hepatitis C viral load by PCR.
17. Clinically significant elevation of GGT (>1.5xULN), bilirubin (>1.25xULN, direct 35%), or INR (>1.2, excluding patients on anti-coagulant therapies) or other clinically significant abnormal laboratory value in the opinion of the investigator.
18. Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 0.
19. Have evidence of serious suicide risk including any history of suicidal behaviour in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, pose a significant suicide risk.
20. Have any concurrent significant medical or psychiatric illness that the investigator considers would make the candidate unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galina Marder, MD, Principal Investigator — Northwell.edu
Locations (1):
- Northwell Health Divison of Rheumatology, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marder G, Quach T, Chadha P, Nandkumar P, Tsang J, Levine T, Schiopu E, Furie R, Davidson A, Narain S. Belimumab treatment of adult idiopathic inflammatory myopathy. Rheumatology (Oxford). 2024 Mar 1;63(3):742-750. doi: 10.1093/rheumatology/kead281. PMID 37326854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 Patients signed consent forms, but two withdrew consent forms before randomization, and were not included in the baseline characteristics analysis, 17 patients were randomized. Two patients out of 17 received less than five doses of Study Drug and as per protocol were excluded from the final efficacy analysis but not safety analysis.
Groups:
- Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase): Patients in this arm will be given belimumab with a background of standard of care therapy during the randomized controlled treatment period.
  Belimumab: Randomized phase: Week 0 - Week 40
  Patients in this arm will continue to receive belimumab during the open label phase of the study (week 40 - week 64)
- Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase): Patients in this arm will be given a placebo with a background of standard of care therapy during the randomized controlled treatment period.
  Placebo: Randomized phase: Week 0 - Week- 40
  Patients in this arm will receive belimumab during the open label phase of the study (week 40 - week 64).
Period: Week 0 - Week 40 (Randomized Phase)
Arm/Group | Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) | Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase)
Started | 10 | 7
Received 5 Doses and Included in Included in the Final Intention-to-treat Analysis | 9 | 6
Completed (9 patients that completed week 16 and were included in 40 week ITT analysis) | 8 | 6
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Period: Week 40 - Week 64 (Open Lable Phase)
Arm/Group | Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) | Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase)
Started | 8 | 6
Completed (all 9 patients that completed week 16 were included in final 64 week ITT analysis.) | 7 | 5
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: 29 screened, 19 enrolled, 2 withdrew consent before randomization. 17 patients started the trial and were randomized. Of 17 patients randomized, 15 received at least 5 doses of belimumab or placebo and were included in the final intention-to-treat analysis. 14 patients (8/9 in the belimumab arm and 6/7 in the placebo arm) completed all 40 weeks of randomized phase. Seven (7/9) patients from belimumab arm and 5 (5/7) from placebo arm completed 24 weeks of open label extension with IV belimumab.
Groups:
- Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase): Patients in this arm will be given a placebo with a background of standard of care therapy during the randomized controlled treatment period.
  Placebo: Randomized phase: Week 0 - Week 40
  Patients in this arm will receive belimumab during the open label phase of the study (week 40 - week 64).
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) | Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase) | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Median (Full Range); unit: years] | 46 [29 to 65] | 52 [33 to 68] | 46 [29 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Subtype of Idiopathic Inflammatory Myositis (IIM) [Count of Participants; unit: Participants]
  Dermatomyositis (DM) | 3 | 3 | 6
  Polymyositis (PM) | 7 | 4 | 11
Disease Duration [Mean (Standard Deviation); unit: years] | 3.5 (3.92) | 4.3 (4.35) | 3.82 (3.99)
Concurrent prednisone (Mean dose (mg)(SD)) [Mean (Standard Deviation); unit: mg] | 7.63 (7.23) | 4.3 (4.5) | 6.25 (6.13)
Percent of participants with concurrent prednisone therapy [Count of Participants; unit: Participants] | 8 | 3 | 11
Percentage of participants on concurrent immunosuppressive agents [Count of Participants; unit: Participants]
  % of participants on Methotrexate or MMF or AZA | 8 | 5 | 13
  % of participants on IVIG | 1 | 6 | 7
  % of participants on Methotrexate or MMF or AZA and IVIG | 4 | 4 | 8
Disease Characteristics Mean (SD) [Mean (Standard Deviation); unit: Score on a scale]
  Manual Muscle Testing (MMT)- measure of muscle strength (0 -150 max muscle strength ) | 115.2 (6.37) | 115.0 (8.25) | 115.12 (10.5)
  Muscle activity score on Visual Analogue Score (0 absence of activity -10 max activity) | 4.54 (1.8) | 5.1 (0.94) | 4.91 (1.58)
  Extra-Muscle activity score Visual Analogue Score (0 - absence of activity -10 max activity) | 0.96 (1.61) | 1.39 (1.36) | 1.10 (1.45)
  Health Assessment Questionnaire (HAQ) disability scale(0 - no disability -3 max disability) | 1.39 (0.68) | 1.2 (0.51) | 1.33 (0.60)
  Myositis Damage Index (MDI) (0 - no damage -10 highest level of damage) | 0.95 (1.52) | 1.7 (2.11) | 1.46 (1.94)

OUTCOME MEASURES:

1. Primary Outcome: Response Rate During Randomized Phase
Description: Definition of Improvement (DOI) is ≥ 20% of improvement in any 3 of the core set measures (CSM) - Manual Muscle Testing, Patient Global , Physician Global, Muscle Enzyme change , HAQ and Extra- muscular activity and no more than 2 CSM worsening by ≥ 25% (excluding MMT).
  Total Improvement Score ( TIS) is a sum of weighted scores of absolute change of core set measures ( MMT, Patient Global , Physician Global, Muscle Enzyme change , HAQ and Extra-muscluar activity ). The scores range from 0 to 100, with higher scores indicating greater improvement. TIS ≥ 40 indicates a moderate response and ≥ 60 TIS indicates a major response.
Time Frame: 40 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase): Patients in this arm will be given a placebo with a background of standard of care therapy during the randomized controlled treatment period.
  Randomized phase_ Week 0 - Week 40
  Patients in this arm will receive belimumab during the open label phase of the study (week 40 - week 64).
- Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase): Patients in this arm will be given belimumab with a background of standard of care therapy during the randomized controlled treatment period.
  Belimumab: Randomized phase: Week 0 - Week 40
  Patients in this arm will continue to receive belimumab during the open label phase of the study (week 40 - week 64)
Arm/Group | Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) | Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase)
Number analyzed (Participants) | 9 | 6
Participants
  Week 40 : Definition of Improvement (DOI) | 3 | 1
  Week 40 : Percent patients reaching Total improvement score of ≥40 | 5 | 2
  Week 40 : Percent of patient with major improvement TIS ≥60 | 2 | 0
Statistical Analysis 1: Comparison: Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) vs Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase); Definition of Improvement (DOI) at week 40; Test type: Superiority; p = 0.60, ANOVA; Risk Ratio (RR) = 0.5, 95% CI 2-sided [0.08 to 2.65]
Statistical Analysis 2: Comparison: Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) vs Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase); Percent patients reaching Total improvement score of ≥40 at Week 40; Test type: Superiority; p = 0.61, ANOVA; Risk Ratio (RR) = 0.6, 95% CI 2-sided [0.16 to 1.82]
Statistical Analysis 3: Comparison: Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) vs Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase); Percent of patient with major improvement TIS ≥60 at Week 40; Test type: Superiority; p = 0.23, ANOVA; Risk Ratio (RR) = 0, 95% CI 2-sided [0 to 1.47]

2. Primary Outcome: Mean Total Improvement Score (TIS) During Randomized Phase
Description: It is a composite measure calculated as a sum of weighted scores assigned to absolute changes for each measure (MMT , Patient Global, Physician Global, Muscle enzymes, Extramuscluar activity and HAQ) . Total score could range from 0 to 100. TIS ≥ 20 indicates minimal improvement, TIS ≥ 40 indicates moderate response and TIS ≥ 60 indicates a major response.
  2016 ACR/EULAR Criteria for Minimal, Moderate, and Major Clinical Response in Adult Dermatomyositis and Polymyositis and Juvenile Dermatomyositis (Aggarwal R et al 2016)
Time Frame: 40 Week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) | Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase)
Number analyzed (Participants) | 9 | 6
score on a scale | 38.8 (24.9) | 37.9 (5.8)
Statistical Analysis 1: Comparison: Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) vs Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase); Mean Total Improvement Score (TIS) during Randomized Phase at Week 40; Test type: Superiority; p = 0.92, ANOVA

3. Secondary Outcome: Response Rate After Open Label Phase
Description: as for outcome 2
Time Frame: 64 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) | Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase)
Number analyzed (Participants) | 9 | 6
Participants
  Week 64 : Definition of Improvement (DOI) | 3 | 0
  Week 64 : Percent patients reaching Total improvement score of ≥40 | 4 | 2
  Week 64 : Percent of patient with major improvement TIS ≥60 | 2 | 0
Statistical Analysis 1: Comparison: Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) vs Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase); Definition of Improvement (DOI) at Week 64; Test type: Superiority; p = 0.23, ANOVA; Risk Ratio (RR) = 0, 95% CI 2-sided [0 to 1.47]
Statistical Analysis 2: Comparison: Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) vs Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase); Percent patients reaching Total improvement score of ≥40 at Week 64; Test type: Superiority; p = 0.99, ANOVA; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.19 to 2.51]
Statistical Analysis 3: Comparison: Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) vs Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase); Percent of patient with major improvement TIS ≥60 at Week 64; Test type: Superiority; p = 0.23, ANOVA; Risk Ratio (RR) = 0, 95% CI 2-sided [0 to 1.47]

4. Secondary Outcome: Mean Total Improvement Score (TIS) After Open Label Phase
Description: Definition of Improvement (DOI) is ≥ 20% of improvement in any 3 of the core set measures (CSM) - Manual Muscle Testing, Patient Global , Physician Global, Muscle Enzyme change , HAQ and Extra- muscular activity and no more than 2 CSM worsening by ≥ 25% (excluding MMT).
  Total Improvement Score ( TIS) is a sum of weighted scores of absolute change of core set measures ( MMT, Patient Global , Physician Global, Muscle Enzyme change , HAQ and Extra-muscluar activity ). The scores range from 0 to 100, with higher scores indicating greater improvement. TIS ≥ 40 indicates a moderate response and ≥ 60 TIS indicates a major response. Minimal, Moderate, and Major Clinical Response in Adult Dermatomyositis and Polymyositis and Juvenile Dermatomyositis (Aggarwal R et al 2016)
Time Frame: 64 Week
Population: In originally assigned Belimumab group 9 patients completed week 16, 8 completed week 40, 7 completed week 64 In originally assigned placebo group 6 patients completed week 16, 6 completed week 40, 5 completed week 64 The response scores at week 40 and 64 were calculated based on number of patients that completed 16 weeks of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) | Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase)
Number analyzed (Participants) | 9 | 6
score on a scale | 41.1 (25.3) | 36 (13.1)
Statistical Analysis 1: Comparison: Arm 1 (Belimumab + SoC (Randomized Phase and Open Label Phase) vs Arm 2 (Placebo + SoC (Randomized Phase) Followed by Belimumab + SoC (Open Label Phase); Mean Total Improvement Score (TIS) after Open Label Phase at 64 Week; Test type: Superiority; p = 0.62, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event information was collected on all enrolled patients from the time of enrollment till last study visit up to 64 weeks.
Groups:
- Arm 1 (Belimumab + SoC (Randomized Phase): Patients in this arm will be given belimumab with a background of standard of care therapy during the randomized controlled treatment period.
  Belimumab: Randomized phase: Week 0 - Week 40
- Arm 2 (Placebo + SoC (Randomized Phase): Patients in this arm will be given a placebo with a background of standard of care therapy during the randomized controlled treatment period.
  Randomized phase_ Week 0 - Week 40
- Open Label Arm 1 and 2 Combined: This is combined group of patients in arm 1 and Arm 2 that were transferred to open label phase and received belimumab with a background of standard of care therapy.
  Belimumab: Randomized phase: Week 40 - Week 64
Arm/Group | Arm 1 (Belimumab + SoC (Randomized Phase) | Arm 2 (Placebo + SoC (Randomized Phase) | Open Label Arm 1 and 2 Combined
All-Cause Mortality (participants affected / at risk) | 6/10 | 6/7 | 6/14
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/7 | 0/14
Other Adverse Events (participants affected / at risk) | 5/10 | 6/7 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Belimumab + SoC (Randomized Phase) (N=10) | Arm 2 (Placebo + SoC (Randomized Phase) (N=7) | Open Label Arm 1 and 2 Combined (N=14)
perforated appendix (Gastrointestinal disorders) | 1 | 0 | NA — perforated appendix
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Belimumab + SoC (Randomized Phase) (N=10) | Arm 2 (Placebo + SoC (Randomized Phase) (N=7) | Open Label Arm 1 and 2 Combined (N=14)
Upper respiratory infection (Infections and infestations) | 2 (2) | 3 (5) | 1 (1) — Upper respiratory infection
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1 — Urinary Tract Infection
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0 — Adjustment disorder
Transaminitis (Hepatobiliary disorders) | 1 | 0 | 0 — Transaminitis
Gout flare (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 | 1 (2)
candida esophagitis (Infections and infestations) | 0 | 0 | 1
fatigue and lightheadedness (General disorders) | 0 | 2 (5) | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT02347891/Prot_SAP_000.pdf